CLINICAL TRIAL: NCT02668328
Title: CGV in Newly Diagnosed Type 2 Diabetes Patients: Effect of Dietary Interventions in the Human Microbiome
Brief Title: Cochlear-Vestibular Ganglion (CVG) in Newly Diagnosed Type 2 Diabetes Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NYUmed
Record Dates: First submitted 2015-12-22; First posted 2016-01-29 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus Type 2 in Obese

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral Intervention (Experimental): The proposed study involves a 2-phase randomized clinical trial in adults with recently diagnosed T2D. Participants will be randomized to a wait-list Control group, BI, or Tailored-BI. In Phase 1, wait-list Control participants will receive 6 months of standard care; BI and Tailored-BI participants will receive 6 months of Active Intervention. In Phase 2, wait-list Control group participants will cross-over to the delayed Tailored-BI, and the BI and Tailored-BI participants will enter a 6-month observation phase to examine maintenance effects of the intervention.
  Interventions: Behavioral: Social Cognitive Theory Tailored Behavioral Intervention

INTERVENTIONS:
Behavioral: Social Cognitive Theory Tailored Behavioral Intervention — The intervention will enhance self-efficacy

SUMMARY:
The proposed study is an integrative scientific undertaking, reflecting the input of experts in the behavioral sciences, mHealth technology, computational biology, endocrinology, biochemistry, and nutrition. The project features a unique translational approach, connecting behavior and biology in an economical manner that provides mechanistic insights into the progression of type 2 diabetes (T2D) and the biologic consequences of behavior change. The project may have profound implications for the clinical management of early T2D.

DETAILED DESCRIPTION:
T2D poses a significant public health problem. Hyperglycemia is associated with a variety of vascular complications, but clinical trials of medication regimes designed to achieve near-normal HbA1c have been mostly negative. The lack of benefit observed in these trials may be due to the fact that they targeted HbA1c rather than glucose variability, and were conducted in patients with established T2D that had already experienced complications of the disease. In early T2D, management of postprandial glycemia may be particularly important for minimization of metabolic memory effects and preservation of beta cell function. Postprandial glycemia in early T2D is largely driven by dietary intake, but research findings that guide clinicians regarding the best dietary approach to prescribe are mixed. Studies done, to-date, have used one-size-fits-all dietary regimes that do not take into consideration the person's unique glycemic response to food. The investigators know from decades of research that behavioral methods are required to engage patients in lifestyle behavior change. The investigators argue that tailoring the approach to the participant's glycemic response and gut microbiome will enhance self-efficacy in ways that cannot be achieved through standard behavioral methods alone and, in turn, reduce glycemic variability and metabolic memory effects.

Co-PI Segal et al. demonstrated that subjects have high between-subject variability in postprandial response to the same food, suggesting that universal dietary recommendations are of limited utility for controlling elevated postprandial glucose. The machine learning algorithm devised by the group integrates multidimensional data to accurately predict personalized postprandial glycemic responses. In a subsequent validation study in 100 participants, they showed that a personally-tailored intervention based on the predicted response resulted in significantly improved postprandial glycemic response, and were accompanied by beneficial changes in gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

* 5 years or less since type 2 diabetes was diagnosed

Exclusion Criteria:

* more 5 years since type 2 diabetes was diagnosed

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Mean Amplitude of Glycemic Excursion (MAGE) | 1 week